CLINICAL TRIAL: NCT00528372
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Dapagliflozin as Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Diet and Exercise
Brief Title: A Phase III Study of BMS-512148 (Dapagliflozin) in Patients With Type 2 Diabetes Who Are Not Well Controlled With Diet and Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-013 LT
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Metformin; Health Services Needs and Demand

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Group 1: Dapagliflozin, 2.5 mg AM (Experimental): Participants with hemoglobin A1c (HbA1c) ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, once each morning for up to 102 weeks.
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Group 1: Dapagliflozin, 10 mg AM (Experimental): Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 10 mg, once each morning for up to 102 weeks.
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Group 1: Dapagliflozin 2.5 mg PM (Experimental): Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, once each evening for up to 102 weeks.
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Group 1: Dapagliflozin, 5 mg PM (Experimental): Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, once each evening for up to 102 weeks.
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Group 1: Dapagliflozin, 10 mg PM (Experimental): Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 10 mg, once each evening for up to 102 weeks.
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Group 2: Dapagliflozin, 5 mg AM (Experimental): Participants with HbA1c ≥10.1% and ≤12% at enrollment received dapagliflozin tablets, 5 mg, once each morning for up to 102 weeks.
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Group 2: Dapagliflozin, 10 mg AM (Experimental): Participants with HbA1c ≥10.1% and ≤12% at enrollment received dapagliflozin tablets, 5 mg, once each morning for up to 102 weeks.
  Interventions: Drug: Dapagliflozin; Drug: Metformin
- Group 1: Dapagliflozin placebo AM & PM (Experimental): Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin placebo once each morning and evening for up to 102 weeks.
  Interventions: Drug: Dapagliflozin placebo; Drug: Metformin
- Group 1: Dapaglifozon, 5 mg AM (Experimental): Participants with (HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, once each morning for up to 102 weeks.
  Interventions: Drug: Dapagliflozin; Drug: Metformin

INTERVENTIONS:
Drug: Dapagliflozin — Tablets; oral; 2.5, 5.0, or 10 mg; once daily in the morning or evening for up to 102 weeks
  Other Names: BMS-512148
  Arms: Group 1: Dapagliflozin 2.5 mg PM; Group 1: Dapagliflozin, 10 mg AM; Group 1: Dapagliflozin, 10 mg PM; Group 1: Dapagliflozin, 2.5 mg AM; Group 1: Dapagliflozin, 5 mg PM; Group 1: Dapaglifozon, 5 mg AM; Group 2: Dapagliflozin, 10 mg AM; Group 2: Dapagliflozin, 5 mg AM
Drug: Dapagliflozin placebo — Tablets, oral, 0 mg, once daily in the morning or evening for up to 102 weeks
  Arms: Group 1: Dapagliflozin placebo AM & PM
Drug: Metformin
  Other Names: Tablets, 500-2000 mg, orally as needed in any arm for rescue, based on protocol specific criteria

SUMMARY:
The purpose of this clinical research study is to determine whether dapagliflozin can improve (decrease) blood glucose values in patients with Type 2 diabetes who have never been treated with medication or have been taking medication for less than 24 weeks since their original diabetes diagnosis. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
All eligible participants will receive single-blind placebo medication during the 2-week lead-in period. All participants may receive additional open-label treatment with metformin, 500-2000 mg, as needed for rescue, based on protocol specific criteria.

ELIGIBILITY:
Key Inclusion Criteria

* Males and females, aged 18 to 77 years
* Type 2 diabetes with inadequate glycemic control, defined as: Group 1, hemoglobin A1c (HbA1c) ≥7% and ≤10%; Group 2, HbA1c ≥10.1% and ≤12.0%
* Drug naive, defined as never having received prescription medications for diabetes, having received prescription medications for diabetes for <24 weeks since the original diagnosis
* C-peptide ≥1.0 ng/mL at enrollment
* Body Mass Index ≤ 45.0 kg/m^2 at enrollment

Key Exclusion Criteria

* Urine albumin:creatinine ratio >1,800 mg/g
* Aspartate aminotransferase >3*upper limit of normal (ULN)
* Alanine aminotransferase >3*ULN
* Serum total bilirubin >2*ULN
* Serum creatinine ≥1.5 mg/dL for men; ≥1.4 mg/dLfor women
* Calcium value outside of the central laboratory normal reference range
* Positive hepatitis B surface antigen
* Positive anti-hepatitis C virus antibody
* Hemoglobin ≤11 g/dL for men; hemoglobin ≤10 g/dL for women
* Creatine kinase >3*ULN
* Abnormal free T4 values
* History of diabetes insipidus
* Symptoms of poorly controlled diabetes, including marked polyuria and polydipsia with greater than 10% weight loss in the 3 months prior to enrollment
* History of diabetic ketoacidosis or hyperosmolar nonketotic coma
* Severe uncontrolled hypertension defined as systolic blood pressure ≥180 mm Hg and/or diastolic blood pressure ≥110 mm Hg
* Any of the following within 6 months of enrollment: Myocardial infarction, cardiac surgery or revascularization, unstable angina, unstable congestive heart failure (CHF), CHF New York Heart Association Class III or IV status, transient ischemic attack or significant cerebrovascular disease, unstable or previously undiagnosed arrhythmia
* History of unstable or rapidly progressing renal disease
* Conditions of congenital renal glucosuria
* Significant hepatic disease, including chronic active hepatitis and/or severe hepatic insufficiency
* Documented history of hepatotoxicity with any medication
* Documented history of severe hepatobiliary disease
* History of hemoglobinopathy, with the exception of sickle cell trait, thalassemia minor, or chronic or recurrent hemolysis
* Donation of blood or blood products to a blood bank, blood transfusion, or participation in a clinical study requiring withdrawal of >400 mL of blood during the 6 weeks prior to enrollment
* Malignancy (with the exception of treated basal cell or treated squamous cell carcinoma) within 5 years of enrollment visit
* Known immunocompromised status, including individuals who had undergone organ transplantation or who had positive HIV results
* Administration of any antidiabetic therapy for more than 14 days (consecutive or not) during the 12 weeks prior to enrollment
* Administration of any antidiabetic therapy, other than any previously specified, at any dose, at any time during the 4 weeks prior to enrollment
* Replacement or chronic systemic corticosteroid therapy, defined as any dose of systemic corticosteroid taken for >4 weeks within 3 months prior to enrollment
* History of bariatric surgery or lap-band procedure
* Administration of sibutramine, phentermine, orlistat, rimonabant, benzphetamine, diethylpropion, methamphetamine, and/or phendimetrazine, within 30 days of enrollment

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1067 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Langkilde, Study Director — AstraZeneca
Locations (71):
- United States (38):
  - 43rd Medical Associates, P.C., Phoenix, Arizona
  - Clin Res Advantage, Inc/East Valley Family Physicians, Plc, Tempe, Arizona
  - Clinical Research Advantage, Inc, Tempe, Arizona
  - Valley Research, Fresno, California
  - Cherlin, Richard, Los Gatos, California
  - Ritchken & First M.D.'S, San Diego, California
  - Torrance Clinical Research, Torrance, California
  - Aurora Family Medicine Center, P.C., Aurora, Colorado
  - Expresscare Clinical Research, Colorado Springs, Colorado
  - Center For Internal Medicine, Denver, Colorado
  - Denver Internal Medicine Group, Denver, Colorado
  - Central Florida Clinical Trials, Altamonte Springs, Florida
  - Family Care Associates, Chipley, Florida
  - Westside Center For Clinical Research, Jacksonville, Florida
  - Panhandle Family Care Associates, Marianna, Florida
  - Louisiana Heart Center, Slidell, Louisiana
  - Jackson, Danny W., Rolling Fork, Mississippi
  - Woodlake Research, Chesterfield, Missouri
  - Nevada Alliance Against Diabetes, Las Vegas, Nevada
  - Slocum-Dickson Medical Group, Pllc, New Hartford, New York
  - Internist Associates Of Central New York, P. C., Syracuse, New York
  - Southgate Medical Group, West Seneca, New York
  - Providence Health Partners, Dayton, Ohio
  - Newark Physician Associates, Newark, Ohio
  - Physician Research, Inc., Zanesville, Ohio
  - Gilbert Medical Research, Llc, Bethany, Oklahoma
  - Integris Family Care Yukon, Yukon, Oklahoma
  - Banksville Medical, Pc, Pittsburgh, Pennsylvania
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Village Family Practice, Houston, Texas
  - Abbott Clinical Research Group, Inc., San Antonio, Texas
  - Sam Clinical Research Center, San Antonio, Texas
  - Taylor/Wade Medical, Bountiful, Utah
  - Optimum Clinical Research, Inc., Salt Lake City, Utah
  - J. Lewis Research, Inc, Salt Lake City, Utah
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - William L. Gray, Md, Spokane, Washington
- Canada (18):
  - Local Institution, Calgary, Alberta
  - Local Institution, Kelowna, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, Moncton, New Brunswick
  - Local Institution, Mount Pearl, Newfoundland and Labrador
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Oakville, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Thornhill, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Drummondville, Quebec
  - Local Institution, Granby, Quebec
  - Local Institution, L'Ancienne-Lorette, Quebec
  - Local Institution, Mirabel, Quebec
  - Local Institution, Saint-Léonard, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Mexico (10):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Durango, Durango
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Guadalajara, Mexico City
  - Local Institution, Mexico, D. F., Mexico City
  - Local Institution, Morelia, Michioacan
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Monterrrey, Nuevo León
  - Local Institution, Mérida, Yucatán
- Russia (5):
  - Local Institution, Kursk
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Smolensk
  - Local Institution, Yaroslaval

REFERENCES:
- [Result] Ferrannini E, Ramos SJ, Salsali A, Tang W, List JF. Dapagliflozin monotherapy in type 2 diabetic patients with inadequate glycemic control by diet and exercise: a randomized, double-blind, placebo-controlled, phase 3 trial. Diabetes Care. 2010 Oct;33(10):2217-24. doi: 10.2337/dc10-0612. Epub 2010 Jun 21. PMID 20566676
- [Result] Bailey CJ, Morales Villegas EC, Woo V, Tang W, Ptaszynska A, List JF. Efficacy and safety of dapagliflozin monotherapy in people with Type 2 diabetes: a randomized double-blind placebo-controlled 102-week trial. Diabet Med. 2015 Apr;32(4):531-41. doi: 10.1111/dme.12624. Epub 2014 Nov 22. PMID 25381876
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Mellander A, Billger M, Johnsson E, Traff AK, Yoshida S, Johnsson K. Hypersensitivity Events, Including Potentially Hypersensitivity-Related Skin Events, with Dapagliflozin in Patients with Type 2 Diabetes Mellitus: A Pooled Analysis. Clin Drug Investig. 2016 Nov;36(11):925-933. doi: 10.1007/s40261-016-0438-3. PMID 27461213
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924
- See also: MB102013_Clinical_Study_Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3672&filename=MB102013_Clinical_Study_Protocol_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1067 participants enrolled, 558 received treatment in the Short-term Period. Of those 558 participants, 469 entered the Long-term Period.
Groups:
- Group 1: Dapagliflozin Placebo: Participants with hemoglobin AIc (HbA1c) ≥7% and ≤10% at enrollment received dapagliflozin placebo once each morning and evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria. During the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 2.5 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria. During the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 5 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria. During the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 10 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 10 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria. During the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 2.5 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, once each evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria. During the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 5 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, once each evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria. During the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 10 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 10 mg, once each evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria. During the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 2: Dapagliflozin, 5 mg AM: Participants with HbA1c ≥10.1% and ≤12% at enrollment received dapagliflozin tablets, 5 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria. During the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 2: Dapagliflozin, 10 mg AM: Participants with HbA1c ≥10.1% and ≤12% at enrollment received dapagliflozin tablets, 10 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria. During the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
Period: Short-term (ST) Period (Day 1-Week 24)
Arm/Group | Group 1: Dapagliflozin Placebo | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM | Group 2: Dapagliflozin, 5 mg AM | Group 2: Dapagliflozin, 10 mg AM
Started | 75 | 65 | 64 | 70 | 67 | 68 | 76 | 34 | 39
Completed | 63 | 60 | 52 | 57 | 58 | 57 | 65 | 28 | 34
Not Completed | 12 | 5 | 12 | 13 | 9 | 11 | 11 | 6 | 5
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 2 | 6 | 0 | 3 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 7 | 1 | 6 | 4 | 6 | 2 | 4
Not completed — Lost to Follow-up | 5 | 1 | 2 | 3 | 3 | 2 | 2 | 3 | 1
Not completed — Poor or noncompliance | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Administration reason by sponsor | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Period: Long-term (LT) Period (Weeks 24-102)
Arm/Group | Group 1: Dapagliflozin Placebo | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM | Group 2: Dapagliflozin, 5 mg AM | Group 2: Dapagliflozin, 10 mg AM
Started | 62 | 59 | 51 | 56 | 58 | 57 | 65 | 28 | 33 (1 patient completed ST phase but withdrew for sponsor administrative reason before start of LT phase)
Completed | 42 | 40 | 43 | 42 | 37 | 42 | 48 | 22 | 27
Not Completed | 20 | 19 | 8 | 14 | 21 | 15 | 17 | 6 | 6
Not completed — Lack of Efficacy | 6 | 6 | 1 | 7 | 7 | 7 | 2 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 1 | 0 | 2 | 3 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 6 | 3 | 3 | 7 | 0 | 4 | 2 | 4
Not completed — Lost to Follow-up | 3 | 2 | 1 | 1 | 0 | 4 | 2 | 3 | 1
Not completed — Poor compliance or noncompliance | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — No longer met study criteria | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Administrative reason by sponsor | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other | 2 | 2 | 1 | 2 | 3 | 0 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants with hemoglobin AIc (HbA1c) concentration ≥7% and ≤10% at enrollment (Group 1) and those with a concentration of HbA1c ≥10.1% and ≤12% at enrollment (Group 2) who received at least 1 dose of study medication.
Groups:
- Group 1: Dapagliflozin Placebo AM & PM: Participants with hemoglobin AIc (HbA1c) ≥7% and ≤10% at enrollment received dapagliflozin placebo once each morning and evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 2.5 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 5 mg AM: Participants with (HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 10 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 10 mg, AM, once each morning for up to 102 weeks.
  Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 2.5 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, once each evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 5 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, once each evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 10 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 10 mg, once each evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 2: Dapagliflozin, 5 mg AM: Participants with HbA1c ≥10.1% and ≤12% at enrollment received dapagliflozin tablets, 5 mg, once each evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 2: Dapagliflozin, 10 mg AM: Participants with HbA1c ≥10.1% and ≤12% at enrollment received dapagliflozin tablets, 10 mg, once each evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Total: Total of all reporting groups
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM | Group 2: Dapagliflozin, 5 mg AM | Group 2: Dapagliflozin, 10 mg AM | Total
Number analyzed (Participants) | 75 | 65 | 64 | 70 | 67 | 68 | 76 | 34 | 39 | 558
Age, Customized [Number; unit: Participants]
  <65 years | 66 | 54 | 54 | 66 | 52 | 53 | 72 | 34 | 36 | 487
  ≥65 and <75 | 8 | 11 | 10 | 4 | 15 | 12 | 4 | 0 | 2 | 66
  ≥75 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 29 | 33 | 36 | 38 | 39 | 37 | 10 | 16 | 282
  Male | 31 | 36 | 31 | 34 | 29 | 29 | 39 | 24 | 23 | 276
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 71 | 63 | 61 | 63 | 65 | 65 | 72 | 31 | 38 | 529
  Black/African American | 2 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 10
  American Indian/Alaskan Native | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 2 | 2 | 1 | 3 | 1 | 0 | 1 | 1 | 1 | 12
  Native Hawaiian/Other Pacific Islanders | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3
  Other | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline to Week 24 in Hemoglobin A1C (HbA1c) (Last Observation Carried Forward [LOCF]): Group 1
Description: HbA1c was measured by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. If no Week 24 assessment was available, the last postbaseline measurement prior to Week 24 was used. For rescued participants, measurements obtained after initiation of rescue medication were not considered in calculating the primary endpoint. Evening dosing groups were summarized as exploratory endpoints.
Time Frame: Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants with nonmissing baseline and Week 24 LOCF values
Measure: Mean (Standard Error); unit: Percent
Groups:
- Group 1: Dapagliflozin, 5 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 10 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 10 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 72 | 64 | 61 | 65 | 62 | 63 | 73
Percent | -0.23 (0.1044) | -0.58 (0.1107) | -0.77 (0.1134) | -0.89 (0.1099) | -0.83 (0.1125) | -0.79 (0.1117) | -0.79 (0.1037)
Statistical Analysis 1: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg AM; Test type: Superiority or Other; p = 0.0207, ANCOVA — Tested at alpha=0.019, applying the Dunnett adjustment; Mean Difference (Final Values) = -0.35, Standard Error of Mean 0.1522
Statistical Analysis 2: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg AM; Test type: Superiority or Other; p = 0.0005, ANCOVA — Tested at alpha=0.019, applying the Dunnett adjustment; Median Difference (Final Values) = -0.54, Standard Error of Mean 0.1541
Statistical Analysis 3: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg AM; Test type: Superiority or Other; p < 0.0001, ANCOVA — Tested at alpha=0.019, applying the Dunnett adjustment; Median Difference (Final Values) = -0.66, Standard Error of Mean 0.1518
Statistical Analysis 4: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg PM; Test type: Superiority or Other; Difference from placebo = -0.61, 95% CI 2-sided [-0.91 to -0.30], Standard Error of Mean 0.1536
Statistical Analysis 5: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg PM; Test type: Superiority or Other; Difference from placebo = -0.56, 95% CI 2-sided [-0.86 to -0.26], Standard Error of Mean 0.1527
Statistical Analysis 6: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg PM; Test type: Superiority or Other; Difference from placebo = -0.56, 95% CI 2-sided [-0.85 to -0.27], Standard Error of Mean 0.1474

2. Secondary Outcome: Adjusted Mean Change From Baseline to Week 24 in Fasting Plasma Glucose Levels (Last Observation Carried Forward [LOCF]): Group 1
Description: Secondary endpoints were tested using a sequential testing procedure and are presented in hierarchical order. Because the primary focus of the entire dapagliflozin program was on morning dosing in a population with HbA1c ≥7% and ≤10%, only data on AM dosing were summarized in secondary efficacy analyses. Data after rescue medication were excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. If no Week 24 assessment was available, glucose levels were recorded from the last postbaseline measurement prior to Week 24. For rescued participants, measurements obtained after initiation of rescue medication was not considered in calculating the endpoint.
Time Frame: Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants with nonmissing baseline and Week 24 LOCF values
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Group 1: Dapagliflozin, 2.5 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, AM, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 5 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, AM, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 75 | 65 | 64 | 70 | 67 | 66 | 73
mg/dL | -4.1 (3.906) | -15.2 (4.196) | -24.1 (4.298) | -28.8 (4.046) | -25.6 (4.132) | -27.3 (4.170) | -29.6 (3.964)
Statistical Analysis 1: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg AM; Test type: Superiority or Other; Sequential testing procedures were used, and no test was performed for this comparison due to the fact that the previous comparison was not significant; Mean Difference (Final Values) = -11.1, Standard Error of Mean 5.734 — Week 24
Statistical Analysis 2: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg AM; Test type: Superiority or Other; p = 0.0007, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -19.9, Standard Error of Mean 5.806 — Week 24
Statistical Analysis 3: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg AM; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistically significant according to hierarchical testing procedure (p<0.05); Mean Difference (Final Values) = -24.7, Standard Error of Mean 5.626 — Week 24
Statistical Analysis 4: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg PM; Test type: Superiority or Other; Difference from placebo = -21.5, 95% CI 2-sided [-32.6 to -10.3], Standard Error of Mean 5.686
Statistical Analysis 5: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg PM; Test type: Superiority or Other; Difference from placebo = -23.3, 95% CI 2-sided [-34.4 to -12.0], Standard Error of Mean 5.711
Statistical Analysis 6: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg PM; Test type: Superiority or Other; Difference from placebo = -25.5, 95% CI 2-sided [-36.4 to -14.5], Standard Error of Mean 5.567

3. Secondary Outcome: Adjusted Mean Change From Baseline to Week 24 in Fasting Plasma Glucose Levels (Last Observation Carried Forward [LOCF]): Group 2
Description: Group 2 was an exploratory group, included to obtain initial efficacy and safety data. No comparator arm was included. Secondary endpoints were tested using a sequential testing procedure and are presented in hierarchical order. Data after rescue medication were excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. If no Week 24 assessment was available, glucose levels were recorded from the last postbaseline measurement prior to Week 24. For rescued participants, measurements obtained after initiation of rescue medication was not considered in calculating the endpoint.
Time Frame: Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants with HbA1c ≥10.1% and ≤12% at enrollment and nonmissing baseline and Week 24 LOCF values
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 2: Dapagliflozin, 5 mg AM | Group 2: Dapagliflozin, 10 mg AM
Number analyzed (Participants) | 25 | 32
mg/dL | -77. (53.39) | -84.3 (61.01)

4. Secondary Outcome: Adjusted Mean Change in Total Body Weight at Week 24 (Last Observation Carried Forward [LOCF]): Group 1
Description: Secondary endpoints were tested using a sequential testing procedure and are presented in hierarchical order. Because the primary focus of the entire dapagliflozin program was on morning dosing in a population with HbA1c ≥7% and ≤10%, only data on AM dosing were summarized. Adjusted mean change from baseline in total body weight at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined). Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: From Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants with nonmissing baseline and Week 24 values
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 75 | 65 | 62 | 69 | 67 | 66 | 74
Kilograms | -2.19 (0.4297) | -3.25 (0.4615) | -2.83 (0.4731) | -3.16 (0.4493) | -3.82 (0.4548) | -3.55 (0.4582) | -3.05 (0.4329)
Statistical Analysis 1: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg AM; Test type: Superiority or Other; [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.06, Standard Error of Mean 0.6307
Statistical Analysis 2: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg AM; Test type: Superiority or Other; p = 0.3101, ANCOVA — Tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -0.65, Standard Error of Mean 0.6388
Statistical Analysis 3: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg AM; Test type: Superiority or Other; p = 0.1189, ANCOVA — Tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -0.97, Standard Error of Mean 0.6223
Statistical Analysis 4: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg PM; Test type: Superiority or Other; Difference from placebo = -1.63, 95% CI 2-sided [-2.86 to -0.41], Standard Error of Mean 0.6254
Statistical Analysis 5: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg PM; Test type: Superiority or Other; Difference from placebo = -1.36, 95% CI 2-sided [-2.60 to -0.13], Standard Error of Mean 0.6279
Statistical Analysis 6: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg PM; Test type: Superiority or Other; Difference from placebo = -0.87, 95% CI 2-sided [-2.06 to 0.33], Standard Error of Mean 0.6103

5. Secondary Outcome: Adjusted Mean Change in Total Body Weight at Week 24 (Last Observation Carried Forward [LOCF]): Group 2
Description: Secondary endpoints were tested using a sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in total body weight at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined). Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was considered an exploratory group, included to obtain initial efficacy and safety data for these patients. No comparator arm was included.
Time Frame: From Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants with HbA1c ≥10.1% and ≤12% at enrollment nonmissing baseline and Week 24 LOCF values.
Measure: Mean (Standard Deviation); unit: Kilograms
Groups:
- Group 2: Dapagliflozin, 5 mg AM: Participants with hemoglobin A1c (HbA1c) ≥10.1% and ≤12% at enrollment received dapagliflozin tablets, 5 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria. During the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
Arm/Group | Group 2: Dapagliflozin, 5 mg AM | Group 2: Dapagliflozin, 10 mg AM
Number analyzed (Participants) | 34 | 37
Kilograms | -2.06 (3.437) | -1.90 (3.539)

6. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose Levels at Week 1 (Last Observation Carried Forward [LOCF]): Group 1
Description: Secondary endpoints were tested using a sequential testing procedure and are presented in hierarchical order. Because the primary focus of the entire dapagliflozin program was on morning dosing in a population with HbA1c ≥7% and ≤10%, only data on AM dosing were summarized. Data after rescue medication was excluded from this analysis. Fasting plasma glucose was measured by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: Baseline to Week 1 (end of Short-term Period)
Population: Randomized participants with nonmissing baseline and Week 24 LOCF values
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 71 | 57 | 56 | 65 | 48 | 54 | 60
mg/dL | -2.4 (2.885) | -2.9 (3.219) | -16.4 (3.248) | -16.1 (3.016) | -14.4 (3.086) | -18.6 (3.219) | -20.3 (3.088)
Statistical Analysis 1: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -0.4, Standard Error of Mean 4.324
Statistical Analysis 2: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -13.9, Standard Error of Mean 4.342
Statistical Analysis 3: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -13.6, Standard Error of Mean 4.176
Statistical Analysis 4: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg PM; Test type: Superiority or Other; Difference from placebo = -12.0, 95% CI 2-sided [-20.3 to -3.7], Standard Error of Mean 4.223
Statistical Analysis 5: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg PM; Test type: Superiority or Other; Difference from placebo = -16.2, 95% CI 2-sided [-24.7 to -7.7], Standard Error of Mean 4.321
Statistical Analysis 6: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg PM; Test type: Superiority or Other; Difference from placebo = -17.9, 95% CI 2-sided [-26.2 to -9.5], Standard Error of Mean 4.228

7. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose Levels at Week 1 (Last Observation Carried Forward [LOCF]): Group 2
Description: as for outcome 6
Time Frame: Baseline to Week 1
Population: Randomized participants with HbA1c ≥10.1% and ≤12% at enrollment with nonmissing baseline and Week 24 LOCF values
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 2: Dapagliflozin, 5 mg AM | Group 2: Dapagliflozin, 10 mg AM
Number analyzed (Participants) | 34 | 37
mg/dL | -54.3 (41.9) | -74.3 (51.09)

8. Secondary Outcome: Adjusted Percentage of Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1c] <7.0%) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using a sequential testing procedure and are presented in hierarchical order. Therapeutic glycemic response is defined as HbA1c <7.0%. Data after rescue medication was excluded from this analysis. If no Week 24 assessment was available, HbA1c was recorded from the last postbaseline measurement prior to Week 24. Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was considered an exploratory group, included to obtain initial efficacy and safety data for these patients. No comparator arm was included. Thus, only key safety and efficacy analyses were performed for Group 2.
Time Frame: Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants who had nonmissing baseline and Week 24 LOCF values
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 72 | 64 | 61 | 65 | 62 | 63 | 73
Percentage of participants | 31.6 | 41.3 | 44.2 | 50.8 | 51.4 | 44.0 | 51.6
Statistical Analysis 1: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg AM; Test type: Superiority or Other; Percentage difference = 9.7
Statistical Analysis 2: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg AM; Test type: Superiority or Other; Percentage difference = 12.6
Statistical Analysis 3: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg AM; Test type: Superiority or Other; Percentage difference = 19.2
Statistical Analysis 4: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg PM; Test type: Superiority or Other; Percent difference from placebo = 19.8, 95% CI 2-sided [4.9 to 34.7]
Statistical Analysis 5: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg PM; Test type: Superiority or Other; Percent difference from placebo = 12.4, 95% CI 2-sided [-2.5 to 27.3]
Statistical Analysis 6: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg PM; Test type: Superiority or Other; Percent difference from placebo = 19.9, 95% CI 2-sided [5.3 to 34.5]

9. Secondary Outcome: Adjusted Mean Change From Baseline to Week 24 in Hemoglobin A1c (HbA1c) in Patients With Baseline HbA1c ≥9.0% (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using a sequential testing procedure and are presented in hierarchical order. If no Week 24 assessment was available, HbA1c was recorded from the last postbaseline measurement prior to Week 24. HbA1c was measured as % of hemoglobin by a central laboratory. The population included randomized patients who received treatment and had baseline HbA1c >9.0%. Data after rescue medication were excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of double-blind study drug. In cases where time of the first dose or assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study drug. Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was considered exploratory, included to obtain initial data. No comparator arm was included. Thus, only key safety and efficacy analyses were performed in Group 2.
Time Frame: Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants with nonmissing baseline and Week24 LOCF values.
Measure: Mean (Standard Error); unit: Percent
Groups:
- Group 1: Dapagliflozin, 2.5 mg AM: Participants with hemoglobin A1c (HbA1c) ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, once each morning for up to 102 weeks.Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapaglifozon, 5 mg AM: Participants with (HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, once each morning for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapaglifozon, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 5 | 8 | 9 | 14 | 11 | 8 | 12
Percent | 0.19 (0.5473) | -1.26 (0.4327) | -2.00 (0.4079) | -2.04 (0.3307) | -1.35 (0.3710) | -1.53 (0.4416) | -1.21 (0.3643)
Statistical Analysis 1: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -1.45, Standard Error of Mean 0.6979
Statistical Analysis 2: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapaglifozon, 5 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -2.19, Standard Error of Mean 0.6828
Statistical Analysis 3: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -2.23, Standard Error of Mean 0.6404
Statistical Analysis 4: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg PM; Test type: Superiority or Other; Difference from placebo = -1.55, 95% CI 2-sided [-3.33 to -0.42], Standard Error of Mean 0.7394
Statistical Analysis 5: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg PM; Test type: Superiority or Other; Difference from placebo = -1.27, 95% CI 2-sided [-2.69 to 0.16], Standard Error of Mean 0.7257
Statistical Analysis 6: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg PM; Test type: Superiority or Other; Difference from placebo = -0.87, 95% CI 2-sided [-2.06 to 0.33], Standard Error of Mean 0.6103

10. Secondary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1c (HbA1c) in Participants With Baseline Body Mass Index (BMI) ≥27 kg/m^2 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using a sequential testing procedure and are presented in hierarchical order. If no Week 24 assessment was available, HbA1c was recorded from the last postbaseline measurement prior to Week 24. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was considered an exploratory group, included to obtain initial efficacy and safety data for these patients. No comparator arm was included. Thus, only key safety and efficacy analyses were performed for Group 2.
Time Frame: Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants with baseline BMI ≥27 kg/m^2 and nonmissing baseline and Week 24 LOCF values
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 58 | 53 | 53 | 59 | 48 | 54 | 60
Percent | -0.21 (0.1210) | -0.58 (0.1265) | -0.73 (0.1267) | -0.88 (0.1201) | -0.81 (0.1329) | -0.76 (0.1255) | -0.80 (0.1194)
Statistical Analysis 1: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -0.37, Standard Error of Mean 0.1750
Statistical Analysis 2: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -0.52, Standard Error of Mean 0.1750
Statistical Analysis 3: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -0.67, Standard Error of Mean 0.1708
Statistical Analysis 4: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg PM; Test type: Superiority or Other; Difference from placebo = -0.60, 95% CI 2-sided [-0.95 to -0.25], Standard Error of Mean 0.1798
Statistical Analysis 5: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg AM; Test type: Superiority or Other; Difference from placebo = -0.55, 95% CI 2-sided [-0.89 to -0.21], Standard Error of Mean 0.1741
Statistical Analysis 6: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg PM; Test type: Superiority or Other; Difference from placebo = -0.58, 95% CI 2-sided [-0.92 to -0.25], Standard Error of Mean 0.1704

11. Secondary Outcome: Adjusted Percentage of Participants Who Achieved Hemoglobin A1c [HbA1c] ≤6.5% (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using a sequential testing procedure and are presented in hierarchical order. If no Week 24 assessment was available, HbA1c was recorded from the last postbaseline measurement prior to Week 24. Data after rescue medication was excluded from this analysis. HbA1c was measured as a percent of hemoglobin. Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was considered an exploratory group, included to obtain initial efficacy and safety data for these patients. No comparator arm was included. Thus, only key safety and efficacy analyses were performed for Group 2.
Time Frame: Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants with HbA1c values at both baseline and Week 24 (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 11 | 17 | 17 | 14 | 62 | 63 | 73
Percentage of participants | 14.5 | 27.2 | 26.6 | 23.1 | 33.4 | 25.8 | 26.0
Statistical Analysis 1: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = 12.6, Standard Error of Mean 6.526
Statistical Analysis 2: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = 12.1, Standard Error of Mean 6.761
Statistical Analysis 3: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = 8.6, Standard Error of Mean 6.334
Statistical Analysis 4: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg PM; Test type: Superiority or Other; Percent difference from placebo = 18.8, 95% CI 2-sided [5.5 to 32.1]
Statistical Analysis 5: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg PM; Test type: Superiority or Other; Percent difference from placebo = 11.3, 95% CI 2-sided [-1.8 to 24.4]
Statistical Analysis 6: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg PM; Test type: Superiority or Other; Percent difference from placebo = 11.4, 95% CI 2-sided [-1.0 to 23.9]

12. Secondary Outcome: Adjusted Mean Change From Baseline to Week 24 in Total Body Weight in Patients With Baseline Body Mass Index ≥27 kg/m^2 (Last Observation Carried Forward)
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in total body weight at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available) was determined. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was considered an exploratory group, included to obtain initial efficacy and safety data for these patients. No comparator arm was included. Thus, only key safety and efficacy analyses were performed for Group 2.
Time Frame: Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants with baseline BMI ≥27 kg/m^2 and nonmissing baseline and Week 24 values
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 60 | 54 | 54 | 63 | 53 | 57 | 61
Kilograms | -2.43 (0.5063) | -3.43 (0.5341) | -2.91 (0.5357) | -3.39 (0.4945) | -4.30 (0.5388) | -3.70 (0.5199) | -3.39 (0.5027)
Statistical Analysis 1: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -1.00, Standard Error of Mean 0.7360
Statistical Analysis 2: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -0.48, Standard Error of Mean 0.7371
Statistical Analysis 3: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg AM; Test type: Superiority or Other; Mean Difference (Final Values) = -0.96, Standard Error of Mean 0.7078
Statistical Analysis 4: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 2.5 mg PM; Test type: Superiority or Other; Difference from placebo = -1.87, 95% CI 2-sided [-3.33 to -0.42], Standard Error of Mean 0.7394
Statistical Analysis 5: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 5 mg PM; Test type: Superiority or Other; Difference from placebo = -1.27, 95% CI 2-sided [-2.69 to 0.16], Standard Error of Mean 0.7257
Statistical Analysis 6: Comparison: Group 1: Dapagliflozin Placebo AM & PM vs Group 1: Dapagliflozin, 10 mg PM; Test type: Superiority or Other; Difference from placebo = -0.97, 95% CI [-2.37 to 0.44], Standard Error of Mean 0.7135

13. Secondary Outcome: Number of Participants With Adverse Events (AE), Hypoglycemia, Related AEs, Death as Outcome, Related Serious AEs (SAEs), SAEs and AEs Leading to Discontinuation, and Hypoglycemia Leading to Discontinuation (Short-term + Long-term Periods)
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or missing relationship to study drug. Includes non-SAEs and hypoglycemia with onset on or after the first date/time of double-blind treatment and on or prior to the last day of short-term plus long-term treatment plus 4 days. Includes SAEs with onset on or after the first date/time of double-blind treatment and on or prior to the last day of short-term plus long-term treatment plus 30 days.
Time Frame: Day 1 to Week 102 (end of Long-term Period) + 30 days
Population: Randomized participants who received at least 1 dose of study medication
Measure: Number; unit: Participants
Groups:
- Group 1: Dapagliflozin Placebo, AM & PM: Participants with hemoglobin AIc (HbA1c) ≥7% and ≤10% at enrollment received dapagliflozin placebo once each morning and evening for up to 102 weeks. In addition, during the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 2.5 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, once each morning for up to 102 weeks. In addition, during the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 5 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, once each morning for up to 102 weeks. In addition, during the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 10 mg AM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 10 mg, once each morning for up to 102 weeks. In addition, during the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 2.5 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, once each evening for up to 102 weeks. In addition, during the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 5 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, once each evening for up to 102 weeks. In addition, during the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
- Group 1: Dapagliflozin, 10 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 10 mg, once each evening for up to 102 weeks. In addition, during the long-term treatment period, participants received metformin, 500 mg, with the morning meal.
Arm/Group | Group 1: Dapagliflozin Placebo, AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM | Group 2: Dapagliflozin, 5 mg AM | Group 2: Dapagliflozin, 10 mg AM
Number analyzed (Participants) | 75 | 65 | 64 | 70 | 67 | 68 | 76 | 34 | 39
Participants
  >=1 AE | 58 | 48 | 43 | 56 | 50 | 50 | 54 | 29 | 33
  >=1 Hypoglycemia | 4 | 3 | 0 | 3 | 2 | 0 | 2 | 1 | 1
  >=1 Related AEs | 15 | 13 | 10 | 17 | 19 | 18 | 21 | 12 | 10
  Deaths | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
  SAEs | 5 | 6 | 4 | 1 | 7 | 5 | 3 | 1 | 0
  >=1 related SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SAEs leading to discontinuation | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0
  AE leading to discontinuation | 4 | 4 | 4 | 5 | 2 | 6 | 7 | 0 | 1
  Hypoglycemia leading to discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Adjusted Mean Change From Baseline to Week 24 in Hemoglobin A1c (HbA1c) (Last Observation Carried Forward [LOCF]): Group 2
Description: HbA1c was measured by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. If no Week 24 assessment was available, the last postbaseline measurement prior to Week 24 was used. For rescued participants, measurements obtained after initiation of rescue medication were not considered in calculating the primary endpoint. Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was considered an exploratory group, included to obtain initial efficacy and safety data for these patients. No comparator arm was included.
Time Frame: Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants with HbA1c ≥10.1% and ≤12% at enrollment and nonmissing baseline and Week 24 LOCF values
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Group 2: Dapagliflozin, 5 mg AM | Group 2: Dapagliflozin, 10 mg AM
Number analyzed (Participants) | 25 | 32
Percent | -2.88 (1.406) | -2.66 (1.261)

15. Secondary Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Marked Laboratory Abnormality (Short-term and Long-term Periods)
Description: Baseline was defined as the last assessment prior to the start of the first dose of the double-blind study medication. Data included from baseline up to and including the last day of treatment plus 4 days. Data after rescue were also included. ULN=upper limit of normal; preRX=pretreatment. Phosphorus, inorganic (high) defined as >=5.6 mg/dL for ages 17-65 years or >=5.1 mg/dL for ages >=66.
Time Frame: Baseline to Week 102 (end of Long-term Period)
Population: Randomized participants who received at least 1 dose of study medication and with laboratory test results available
Measure: Number; unit: Participants
Groups:
- Group 1: Dapagliflozin Placebo: Participants with hemoglobin AIc (HbA1c) ≥7% and ≤10% at enrollment received dapagliflozin placebo once each morning and evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 2.5 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 2.5 mg, PM, once each evening for up to 102 weeks.
  Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 5 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 5 mg, PM, once each evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
- Group 1: Dapagliflozin, 10 mg PM: Participants with HbA1c ≥7% and ≤10% at enrollment received dapagliflozin tablets, 10 mg, PM, once each evening for up to 102 weeks. Participants also received metformin tablets, 500-2000 mg, orally as needed for rescue based on protocol specific criteria.
Arm/Group | Group 1: Dapagliflozin Placebo | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM | Group 2: Dapagliflozin, 5 mg AM | Group 2: Dapagliflozin, 10 mg AM
Number analyzed (Participants) | 75 | 65 | 62 | 70 | 67 | 66 | 73 | 34 | 39
Participants
  Hematocrit (>55%) | 0 | 1 | 0 | 2 | 2 | 1 | 4 | 2 | 4
  Hematocrit (>60%) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Hemoglobin (>18 g/dL) | 0 | 3 | 2 | 4 | 2 | 1 | 6 | 3 | 5
  Glucose ( >350 mg/dL) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose (<54 mg/dL) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Creatine kinase (>5*ULN) | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0
  Creatine kinase (>10*ULN) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
  Calcium, total (<7.5 mg/dL) | 3 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0
  Bicarbonate (<=13 mEq/L) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, serum (>=6 mEqL) | 3 | 1 | 1 | 2 | 4 | 1 | 1 | 1 | 1
  Sodium, serum (<130 mEq/L) | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Sodium, serum (>150 mEq/L) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Phosphorus, inorganic (high) | 2 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 2
  Albumin/creatinine ratio (>1800 mg/g) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine (>=1.5 preRX creatinine) | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1

16. Secondary Outcome: Number of Participants With Elevated Levels of Liver Enzymes on Laboratory Test Results (Short-term and Long-term Periods)
Description: Data after rescue was included. AST=aspartate aminotransferase; ALT=alanine aminotransferase; ALP=alkaline phosphatase. Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was considered an exploratory group, included to obtain initial efficacy and safety data for these patients. No comparator arm was included. Thus, only key safety and efficacy analyses were performed for Group 2.
Time Frame: Day 1 to Week 102 (end of Long-term Period)
Population: Randomized participants who received at least 1 dose of study medication and with laboratory test results available
Measure: Number; unit: Participants
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 75 | 65 | 64 | 70 | 67 | 68 | 76
Participants
  AST >3*ULN (n=75, 65, 62, 70, 67, 67, 74, 34, 37)) | 0 | 1 | 1 | 0 | 5 | 1 | 4
  AST >5*ULN (n=75, 65, 62, 70, 67, 67, 74) | 0 | 0 | 0 | 0 | 2 | 0 | 0
  ALT >3*ULN (n=75, 65, 62, 70, 67, 67, 74) | 1 | 1 | 2 | 1 | 0 | 0 | 0
  ALT >5*ULN (n=75, 65, 62, 70, 67, 67, 74) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Bilirubin >1.5 ULN (n=75, 65, 62, 70, 67, 67, 74) | 2 | 0 | 1 | 0 | 2 | 1 | 0
  Bilirubin >2*ULN (n=75, 65, 62, 70, 67, 67, 74) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ALP >1.5*ULN (n=75, 65, 62, 70, 67, 67, 74) | 4 | 3 | 1 | 1 | 4 | 3 | 2

17. Secondary Outcome: Number of Participants With Changes From Baseline in Electrocardiogram (ECG) Findings (Last Observation Carried Forward {LOCF])
Description: 12-Lead ECGs were performed at entry into lead-in period Day -7 visit and Week 24/end of treatment visit (LOCF) on participants who were supine. ECGs were assessed by the investigator. Baseline was Day -7 for this parameter, and data after rescue were included.The Week 102 value is the last observation, regardless of rescue prior to Week 102 if no Week 102 measurement was available. Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was considered an exploratory group, included to obtain initial efficacy and safety data for these patients. No comparator arm was included. Thus, only key safety and efficacy analyses were performed for Group 2.
Time Frame: Baseline to Week 24 (end of Short-term Period)
Population: Randomized participants who received at least 1 dose of study medication and who had measurements available
Measure: Number; unit: Participants
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Number analyzed (Participants) | 75 | 65 | 64 | 70 | 67 | 68 | 76
Participants
  Baseline: Normal/Week 24: Normal | 38 | 36 | 32 | 31 | 33 | 33 | 35
  Baseline: Normal/Week 24: Abnormal | 6 | 3 | 5 | 1 | 3 | 6 | 10
  Baseline: Normal/Week 24: Not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Abnormal/Week 24: Normal | 5 | 2 | 3 | 6 | 4 | 4 | 10
  Baseline: Abnormal/Week 24: Abnormal | 18 | 17 | 11 | 17 | 17 | 14 | 11
  Baseline: Abnormal/Week 24: Not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Not reported/Week 24: Normal | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basline: Not reported/Week 24: Abnormal | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: Not reported/Week 24: Not reported | 8 | 7 | 13 | 15 | 10 | 11 | 10

ADVERSE EVENTS:
Time Frame: Day 1 to Week 102 (end of Long-term Period)
Description: Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was considered an exploratory group, included to obtain initial efficacy and safety data for these patients. No comparator arm was included.
Arm/Group | Group 1: Dapagliflozin Placebo AM & PM | Group 1: Dapagliflozin, 2.5 mg AM | Group 1: Dapagliflozin, 5 mg AM | Group 1: Dapagliflozin, 10 mg AM | Group 1: Dapagliflozin, 2.5 mg PM | Group 1: Dapagliflozin, 5 mg PM | Group 1: Dapagliflozin, 10 mg PM
Serious Adverse Events (participants affected / at risk) | 5/75 | 6/65 | 4/64 | 1/70 | 7/67 | 5/68 | 3/76
Other Adverse Events (participants affected / at risk) | 40/75 | 40/65 | 33/64 | 41/70 | 38/67 | 39/68 | 39/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Dapagliflozin Placebo AM & PM (N=75) | Group 1: Dapagliflozin, 2.5 mg AM (N=65) | Group 1: Dapagliflozin, 5 mg AM (N=64) | Group 1: Dapagliflozin, 10 mg AM (N=70) | Group 1: Dapagliflozin, 2.5 mg PM (N=67) | Group 1: Dapagliflozin, 5 mg PM (N=68) | Group 1: Dapagliflozin, 10 mg PM (N=76)
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Albumin urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Glomerulonephritis acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malacoplakia vesicae (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine albumin/creatinine ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Dapagliflozin Placebo AM & PM (N=75) | Group 1: Dapagliflozin, 2.5 mg AM (N=65) | Group 1: Dapagliflozin, 5 mg AM (N=64) | Group 1: Dapagliflozin, 10 mg AM (N=70) | Group 1: Dapagliflozin, 2.5 mg PM (N=67) | Group 1: Dapagliflozin, 5 mg PM (N=68) | Group 1: Dapagliflozin, 10 mg PM (N=76)
Bronchitis (Infections and infestations) | 5 | 2 | 1 | 4 | 5 | 4 | 4
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 4 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 2 | 4 | 4 | 7 | 6
Influenza (Infections and infestations) | 3 | 7 | 5 | 5 | 1 | 6 | 5
Pharyngitis (Infections and infestations) | 6 | 1 | 6 | 5 | 6 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 1 | 5 | 3 | 2 | 9
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 6 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 4 | 5 | 2 | 6 | 7
Dizziness (Nervous system disorders) | 2 | 3 | 1 | 2 | 6 | 4 | 3
Hypertension (Vascular disorders) | 3 | 4 | 4 | 3 | 5 | 3 | 4
Oedema peripheral (General disorders) | 2 | 1 | 2 | 1 | 2 | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 3 | 3 | 2 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 5 | 6 | 3 | 8 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 2 | 4 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 1 | 1 | 3 | 4
Urinary tract infection (Infections and infestations) | 3 | 3 | 5 | 5 | 4 | 7 | 5
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 4 | 2 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 4
Toothache (Gastrointestinal disorders) | 0 | 4 | 0 | 1 | 4 | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 2 | 1 | 2 | 1 | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 3 | 3 | 3 | 3 | 3
Gastritis (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 2 | 3 | 4
Headache (Nervous system disorders) | 9 | 6 | 5 | 6 | 4 | 11 | 10
Nasopharyngitis (Infections and infestations) | 7 | 11 | 5 | 10 | 11 | 9 | 7

LIMITATIONS AND CAVEATS:
Group 2 (patients with enrollment baseline HbA1c >10% and ≤2%) was an exploratory group, included to obtain initial efficacy and safety data. No comparator arm was included. Thus, only key safety and efficacy analyses were performed for Group 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.